CLINICAL TRIAL: NCT06206200
Title: The Effects of Cognitive Dual-Tasking in Later Stages of Rehabilitation After ACL Reconstruction
Acronym: AMIRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2023-0365
Record Dates: First submitted 2024-01-02; First posted 2024-01-16 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Athrogenic Muscle Responses; ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual task training (Experimental): Patients will recieve 12 sessions (2x/week) of standard of care exercise-based physiotherapy with implementation of cognitive dual task training. This implies that the patients will perform cognitive tasks simultaneously during at least 50% of their physical rehabilitative exercises.
  Interventions: Other: Cognitive dual task training (intervention group)
- Standard of care physiotherapy (Active Comparator): Patients will recieve 12 sessions (2x/week) of standard of care exercise-based physiotherapy without implementation of cognitive dual task training.
  Interventions: Other: Standard of care physiotherapy (control group)

INTERVENTIONS:
Other: Cognitive dual task training (intervention group) — Simultaneously performing cognitive tasks and motor rehabilitative exercises.
  Arms: Dual task training
Other: Standard of care physiotherapy (control group) — The current best physical therapy treatment for patients with anterior cruciate ligament reconstruction based on existing scientific evidence.
  Arms: Standard of care physiotherapy

SUMMARY:
Anterior cruciate ligament (ACL) injuries are common in sports and often require a long and challenging rehabilitation process. Athletes who sustain these injuries typically engage in pivoting and cutting sports, where these motor tasks must be performed simultaneously with cognitive tasks such as decision-making and keeping an eye on the opponent. Directing attention to both cognitive and motor tasks leads to cognitive-motor interference, which is associated with movement patterns that increase the risk of ACL (re)injury.

Therefore, it is crucial that before returning to such demanding sports after ACL reconstruction, athletes sufficiently develop and automate safe yet efficient motor skills to free up attentional capacity for decision-making, thereby reducing the risk of suboptimal movement patterns and reinjury.

However, current rehabilitation programs often primarily focus on the motor component in a single-task manner, giving insufficient attention to the cognitive component that is inseparable from sports.

This randomized controlled trial aims to investigate the effects of implementing motor-cognitive dual tasks in the end phase rehabilitation after ACL reconstruction on muscle function, functional outcomes, and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old.
* Having suffered an ACL rupture.
* Undergoing a surgical ACL reconstruction in the AZ Delta hospital in Roeselare (Campus Brugsesteenweg).

Exclusion Criteria:

* Revision ACL reconstruction.
* Other severe injuries to the lower limbs within the past year.
* Muscle or neurological disorders affecting lower limb functioning.
* Fibromyalgia or chronic fatigue syndrome.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Psychological readiness to return to sport | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Questioned using the ACL-RSI. Scores range from 0 to 100. Higher scores indicate higher psychological readiness.
Quadriceps and hamstrings activity / cocontraction during hop tasks | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Electromyographical measurement of quadriceps and hamstrings activation during hop tasks.
Patient reported knee function | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Questioned using the Knee Injury and Osteoarthritis Outcome Score (KOOS) with its different subscores. Scores on the KOOS range from 0-100, with 0 representing the greatest possible problems in terms of knee function and 100 representing no problems.
Jumping height in hop tests | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Performance in single hop tests and a single leg drop-jump expressed by jump height in centimeters.
Activity level | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Questioned using the Tegner Score. The scores range from 0 to 10, with higher scores indicating higher activity levels.
Voluntary quadriceps activation | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  A force-based isometric biodex measurement using the interpolated twitch/superimposed burst technique.

SECONDARY OUTCOMES:
Quadriceps and hamstrings strength | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Measured on the biodex.
Kinesiophobia | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Questioned using the Tampa Scale of Kinesiophobia (TSK). Scores on the TSK range from 17 to 68, with higher scores indicating more kinesiophobia.
Subjective knee stability | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Questioned using the first question of the Lysholm questionnaire. Scores range from 0 to 25 with 25 indicating no symptoms of subjective instability.
The amount of pain that the subjects experience. | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Questioned using a Numeric Rating Scale. The scores range between 0 and 10 with 10 0representing the highest level of pain.

OTHER OUTCOMES:
Duration of ground contact in hop tests | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Performance in single hop tests and a single leg drop-jump expressed by the duration of ground contact.
Performance in the T-agility test | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  It will be measured how much time subjects require to complete a T-agility test.
Strength endurance during timed single leg step down and timed single leg squat | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  The strength endurance of the subjects will be evaluated by the amount of repetitions they can perform in a time span of 30 seconds.
Expectations regarding return to sport | 5 months post ACL reconstruction (= prior to intervention); 7 months post ACL reconstruction (= after the intervention); 9 months post ACL reconstruction (= after a 2 month retention period)
  Questioned using the Tegner Score: 'how active do you want to be at the end of your rehabilitation?'. The scores range from 0 to 10, with higher scores indicating higher activity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Delta Roeselare (Campus Brugsesteenweg), Roeselare, West-Vlaanderen, Belgium